CLINICAL TRIAL: NCT01904500
Title: Peri-operative Cefazolin Prophylaxis at Time of Cesarean Delivery in the Obese Gravida
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Omar M Young, MD, Clinical Fellow, Division of Maternal-Fetal Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO13040497
Record Dates: First submitted 2013-07-10; First posted 2013-07-22 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Pregnancy
Keywords: Cesarean delivery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Cefazolin 2 grams (Other)
  Interventions: Drug: Pre-operative cefazolin
- Cefazolin 3 grams (Active Comparator)
  Interventions: Drug: Pre-operative cefazolin

INTERVENTIONS:
Drug: Pre-operative cefazolin

SUMMARY:
Obesity has become an increasingly prevalent public health problem in the United States, reaching epidemic proportions. According to 2009 CDC epidemiologic data on obesity in the United States, 35.7% of the United States population is considered overweight or obese. Currently, on the review of the literature, over 20% of pregnancies in this country are complicated by maternal obesity. Obesity has been well demonstrated to be correlated with numerous adverse pregnancy outcomes such hypertensive disorders of pregnancy, gestational diabetes, and increased rates of operative delivery. Moreover, obesity, irrespective of pregnancy, has been demonstrated to be an independent risk factor for the development of postoperative surgical site infections. Development of such infections can have both consequential long-term medical sequelae for patients and economic impacts on the health care system at large. Cefazolin, a first generation hydrophilic cephalosporin whose clearance is exclusively mediated via the kidneys unchanged, is used as pre-operative antibiotic prophylaxis for cesarean deliveries. The current accepted standard of care is to administer 2 grams of cefazolin within 60 minutes of skin incision. Studies of drug concentrations of cephalosporins for pre-operative antibiotic prophylaxis in obese bariatric patients have shown that therapeutic concentrations may not be achieved in both tissue and plasma. Limited data exist in pregnancy. Therefore, it is the goal of this study to investigate whether obese patients presenting for cesarean delivery require an increased dosing amount of pre-operative antibiotic prophylaxis. This study will randomized women with a pre-pregnancy body mass index of 30 kg/m2 or more who are presenting for their scheduled cesarean delivery to receive either 2 grams or 3 grams of cefazolin for pre-operative antibiotic prophylaxis. By drawing blood at specific time points in the peri-operative period and extracting adipose tissue samples during cesarean delivery, this study will investigate the pharmacokinetics of cefazolin in both the plasma and tissues of the obese gravida.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than 30kg/m2
* Those women having scheduled primary or repeat cesarean delivery

Exclusion Criteria:

* Type 1 and Type 2 Insulin Dependent Diabetes Mellitus
* Autoimmune disease, including systemic lupus erythematosus
* History of chronic renal disease
* Those using chronic corticosteroids
* Those with a history of a previous wound breakdown
* Those who have an allergy to cephalosporins whose reaction includes anaphylaxis, urticaria or other systemic consequences
* Those who are unable to receive their antibiotics in a timely fashion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Plasma area under the curve (AUC) of cefazolin | Within the first 8 hours after skin incision
  The primary aim of this study will be to evaluate the plasma area under the curve (AUC) of cefazolin in both the 2 grams and 3 grams groups. Blood samples will be obtained prior to administration of cefazolin and then 15 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 4 hours, 6 hours and 8 hours from administration of cefazolin

SECONDARY OUTCOMES:
Adipose tissue concentrations of cefazolin | Adipose tissue samples will be assessed at time of skin incision, hysterotomy closure and then fascial closure.
Cmax | Within the first 8 hours after skin incision
Drug Clearance (Cl) | Within the first 8 hours after skin incision
Volume of distribution (Vd) | Within the first 8 hours after skin incision
Absolute drug concentrations in plasma and tissue | Within the first 8 hours after skin incision
Tissue to Plasma (T/P) Drug Concentration Ratios | Within the first 8 hours after skin incision
Surgical site infection fo any type | Participants will be followed for the duration of their hospital stay and will be called at 6 weeks from surgery
Cord blood concentration | At time of delivery
Urine drug concentration | 8 hours
  Samples to be obtained up to 8 hours post cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Omar Young, MD, Principal Investigator — Clinical Fellow, Division of Maternal-Fetal Medicine
Locations (1):
- Magee-Women's Hospital/University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity in the United States, 2009-2010. NCHS Data Brief. 2012 Jan;(82):1-8. PMID 22617494
- [Background] ACOG Practice Bulletin No. 120: Use of prophylactic antibiotics in labor and delivery. Obstet Gynecol. 2011 Jun;117(6):1472-1483. doi: 10.1097/AOG.0b013e3182238c31. No abstract available. PMID 21606770
- [Background] Dinsmoor MJ, Gilbert S, Landon MB, Rouse DJ, Spong CY, Varner MW, Caritis SN, Wapner RJ, Sorokin Y, Miodovnik M, O'Sullivan MJ, Sibai BM, Langer O; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Perioperative antibiotic prophylaxis for nonlaboring cesarean delivery. Obstet Gynecol. 2009 Oct;114(4):752-756. doi: 10.1097/AOG.0b013e3181b8f28f. PMID 19888031
- [Background] Pai MP, Bearden DT. Antimicrobial dosing considerations in obese adult patients. Pharmacotherapy. 2007 Aug;27(8):1081-91. doi: 10.1592/phco.27.8.1081. PMID 17655508
- [Background] Pevzner L, Swank M, Krepel C, Wing DA, Chan K, Edmiston CE Jr. Effects of maternal obesity on tissue concentrations of prophylactic cefazolin during cesarean delivery. Obstet Gynecol. 2011 Apr;117(4):877-882. doi: 10.1097/AOG.0b013e31820b95e4. PMID 21422859
- [Background] Craig WA. Interrelationship between pharmacokinetics and pharmacodynamics in determining dosage regimens for broad-spectrum cephalosporins. Diagn Microbiol Infect Dis. 1995 May-Jun;22(1-2):89-96. doi: 10.1016/0732-8893(95)00053-d. PMID 7587056
- [Background] Tita ATN, Rouse DJ, Blackwell S, Saade GR, Spong CY, Andrews WW. Emerging concepts in antibiotic prophylaxis for cesarean delivery: a systematic review. Obstet Gynecol. 2009 Mar;113(3):675-682. doi: 10.1097/AOG.0b013e318197c3b6. PMID 19300334
- [Background] Ho VP, Nicolau DP, Dakin GF, Pomp A, Rich BS, Towe CW, Barie PS. Cefazolin dosing for surgical prophylaxis in morbidly obese patients. Surg Infect (Larchmt). 2012 Feb;13(1):33-7. doi: 10.1089/sur.2010.097. Epub 2012 Feb 8. PMID 22316145
- [Background] van Kralingen S, Taks M, Diepstraten J, van de Garde EM, van Dongen EP, Wiezer MJ, van Ramshorst B, Vlaminckx B, Deneer VH, Knibbe CA. Pharmacokinetics and protein binding of cefazolin in morbidly obese patients. Eur J Clin Pharmacol. 2011 Oct;67(10):985-92. doi: 10.1007/s00228-011-1048-x. Epub 2011 Apr 16. PMID 21499760
- [Background] Toma O, Suntrup P, Stefanescu A, London A, Mutch M, Kharasch E. Pharmacokinetics and tissue penetration of cefoxitin in obesity: implications for risk of surgical site infection. Anesth Analg. 2011 Oct;113(4):730-7. doi: 10.1213/ANE.0b013e31821fff74. Epub 2011 Jun 3. PMID 21642605
- [Background] Liu P, Derendorf H. Antimicrobial tissue concentrations. Infect Dis Clin North Am. 2003 Sep;17(3):599-613. doi: 10.1016/s0891-5520(03)00060-6. PMID 14711079
- [Background] Forse RA, Karam B, MacLean LD, Christou NV. Antibiotic prophylaxis for surgery in morbidly obese patients. Surgery. 1989 Oct;106(4):750-6; discussion 756-7. PMID 2799651
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Allegaert K, van Mieghem T, Verbesselt R, de Hoon J, Rayyan M, Devlieger R, Deprest J, Anderson BJ. Cefazolin pharmacokinetics in maternal plasma and amniotic fluid during pregnancy. Am J Obstet Gynecol. 2009 Feb;200(2):170.e1-7. doi: 10.1016/j.ajog.2008.08.067. Epub 2008 Nov 11. PMID 19006783
- [Background] Philipson A, Stiernstedt G, Ehrnebo M. Comparison of the pharmacokinetics of cephradine and cefazolin in pregnant and non-pregnant women. Clin Pharmacokinet. 1987 Feb;12(2):136-44. doi: 10.2165/00003088-198712020-00004. PMID 3829560
- [Background] Kato Y, Takahara S, Kato S, Kubo Y, Sai Y, Tamai I, Yabuuchi H, Tsuji A. Involvement of multidrug resistance-associated protein 2 (Abcc2) in molecular weight-dependent biliary excretion of beta-lactam antibiotics. Drug Metab Dispos. 2008 Jun;36(6):1088-96. doi: 10.1124/dmd.107.019125. Epub 2008 Mar 13. PMID 18339814
- [Background] Sakurai Y, Motohashi H, Ogasawara K, Terada T, Masuda S, Katsura T, Mori N, Matsuura M, Doi T, Fukatsu A, Inui K. Pharmacokinetic significance of renal OAT3 (SLC22A8) for anionic drug elimination in patients with mesangial proliferative glomerulonephritis. Pharm Res. 2005 Dec;22(12):2016-22. doi: 10.1007/s11095-005-8383-5. Epub 2005 Nov 1. PMID 16247710